CLINICAL TRIAL: NCT00428116
Title: Optimizing Pediatric HIV-1 Treatment, Nairobi, Kenya (0-4.5 Month Randomized Controlled Trial)
Brief Title: Optimizing Pediatric HIV-1 Treatment, Nairobi, Kenya
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommended termination because TI was safe but not durable.
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Nairobi (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001675; R01HD023412 (NIH)
Record Dates: First submitted 2007-01-22; First posted 2007-01-29 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Pediatric; HAART; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interrupted HAART (No Intervention): After 24 months of treatment with HAART, half the eligible infants will be randomized to interrupted treatment and followed for 18 months.
- Continued HAART (Active Comparator): After 24 months of treatment with HAART, half the eligible infants will be randomized to continued treatment with HAART for 18 months.
  Interventions: Drug: HAART

INTERVENTIONS:
Drug: HAART — Combination first line antiretrovirals as previously described.
  Arms: Continued HAART

SUMMARY:
Given the high mortality associated with infant HIV-1 and the fact that surrogate markers are poorly predictive of mortality risk,empiric highly active antiretroviral therapy (HAART) initiation is started in infants younger than 12 months. A problem with this approach is that it obligates infants to life-long therapy, which may be associated with cumulative drug toxicity, poor adherence, and treatment failure. Early HAART for prevention of mortality during the first 2 years of life has potential to salvage immune function and alter viral set-point, allowing withdrawal of therapy, perhaps for several years, until subsequent CD4% decline requires it. This untested approach is attractive because it combines the survival benefits of early pediatric HAART therapy with the benefits of antiretroviral deferral.

One hundred and fifty infants who initiated HAART at <13 months of age will be treated with HAART regimen for 24 months after which those who have immune reconstitution and adequate growth (~100) will be randomized to continued versus deferred therapy. Clinical outcomes, growth, and toxicity will be compared in these children to determine if interruption is a safe and beneficial strategy. Follow-up in this studies will be closely monitored by an external Data Safety and Monitoring Board (DSMB).

DETAILED DESCRIPTION:
Hypothesis: Deferring antiretroviral therapy in infants who have immune reconstitution and adequate growth following early therapy of primary infection (initiated HAART during primary infection at less than 13 months of age) will not compromise clinical status or growth and may spare antiretroviral toxicity.

Specific Aim/Primary Objective: To compare growth and morbidity in infants (who initiated HAART during primary infection at less than or equal to 13 months of age with subsequently normalized CD4% and growth following 24 months of HAART) randomized to deferred versus continuous therapy and followed for an additional 18 months.

Secondary Aim/Secondary Objective: To determine predictors of non-progression of HIV among the infants, including: age, adherence, HIV-1 specific immune responses, baseline HIV-1 RNA, CD4 percent and immune activation.

Design: Randomized clinical trial involving HIV-1 treatment of infants (<13 months old) for 24 months, followed by randomization and 18 months follow-up of children randomized to continued versus deferred treatment. This trial is unblinded.

Population: HIV-1 infected infants (<13 months) newly initiating HAART and HIV-1 infected infants already receiving HAART who initiated HAART at age <13 months will be enrolled. After 24 months of treatment follow-up, children with CD4% > 25% and normalized growth will be retained in the study and randomized.

Sample size: 150 infants will be enrolled of which 100 are expected to be eligible for randomization (50 in each arm).

Treatment: All infants will be treated with HAART according to WHO and Kenyan national guidelines. The specific regimens that will be used as a part of this study are:

First line regimen

* AZT/3TC/NVP (zidovudine/lamivudine/nevirapine)
* d4T/3TC/NVP (stavudine/lamivudine/nevirapine)
* AZT/3TC/ABC (zidovudine/lamivudine/abacavir)
* d4T/3TC/ABC (stavudine/lamivudine/abacavir)
* ABC/3TC/NVP (abacavir/lamivudine/nevirapine)

Second line regimen - ddI/ABC/LPV/r (didanosine/abacavir/lopinavir-ritonavir (Kaletra))

For infants with prior exposure to nevirapine as part of PMTCT:

First line regimen

- AZT/3TC/LPV/r (zidovudine/lamivudine/lopinavir-ritonavir (kaletra))

ELIGIBILITY:
Inclusion Criteria:

A. Infants newly initiating HAART

* Less than 13 months of age
* HIV-1 DNA detection with confirmation (positive on two HIV-1 DNA filter paper tests)
* Caregiver of infant plans to reside in Nairobi for at least 3 years (reported by caregiver)
* Caregiver is able to provide sufficient location information

B. Infants already receiving HAART

* Initiated HAART at <13 months of age
* Records confirming HIV positive status
* Documentation of CD4% and weight prior to HAART initiation
* Must be on 1st line drug regimen

Eligibility for randomization:

* Completed 24 months of treatment with HAART
* Normalized growth: weight for height z-score (WHZ) > -0.5; Child's weight must be above the 5th weight-for-age percentile and the weight curve must not be flat or falling (i.e. cross 2 major percentile lines or more over the past 3 months)
* CD4% > 25
* Children who recently initiated or who require anti-tuberculosis treatment at the time of randomization will be ineligible for randomization.

Max Age: 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2007-09; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Wamalwa, MMed, MPH, Principal Investigator — Department of Paediatrics and Child Health, Kenyatta National Hospital, University of Nairobi; Grace C John-Stewart, MD, PhD, Principal Investigator — University of Washington

REFERENCES:
- [Result] Wamalwa D, Benki-Nugent S, Langat A, Tapia K, Ngugi E, Moraa H, Maleche-Obimbo E, Otieno V, Inwani I, Richardson BA, Chohan B, Overbaugh J, John-Stewart GC. Treatment interruption after 2-year antiretroviral treatment initiated during acute/early HIV in infancy. AIDS. 2016 Sep 24;30(15):2303-13. doi: 10.1097/QAD.0000000000001158. PMID 27177316
- [Result] Njuguna IN, Wagner AD, Cranmer LM, Otieno VO, Onyango JA, Chebet DJ, Okinyi HM, Benki-Nugent S, Maleche-Obimbo E, Slyker JA, John-Stewart GC, Wamalwa DC. Hospitalized Children Reveal Health Systems Gaps in the Mother-Child HIV Care Cascade in Kenya. AIDS Patient Care STDS. 2016 Mar;30(3):119-24. doi: 10.1089/apc.2015.0239. PMID 27308805
- [Result] Sridharan G, Wamalwa D, John-Stewart G, Tapia K, Langat A, Moraa Okinyi H, Adhiambo J, Chebet D, Maleche-Obimbo E, Karr CJ, Benki-Nugent S. High Viremia and Wasting Before Antiretroviral Therapy Are Associated With Pneumonia in Early-Treated HIV-Infected Kenyan Infants. J Pediatric Infect Dis Soc. 2017 Sep 1;6(3):245-252. doi: 10.1093/jpids/piw038. PMID 27481854
- [Result] Asbjornsdottir KH, Hughes JP, Wamalwa D, Langat A, Slyker JA, Okinyi HM, Overbaugh J, Benki-Nugent S, Tapia K, Maleche-Obimbo E, Rowhani-Rahbar A, John-Stewart G. Differences in virologic and immunologic response to antiretroviral therapy among HIV-1-infected infants and children. AIDS. 2016 Nov 28;30(18):2835-2843. doi: 10.1097/QAD.0000000000001244. PMID 27603293
- [Result] Wagner A, Slyker J, Langat A, Inwani I, Adhiambo J, Benki-Nugent S, Tapia K, Njuguna I, Wamalwa D, John-Stewart G. High mortality in HIV-infected children diagnosed in hospital underscores need for faster diagnostic turnaround time in prevention of mother-to-child transmission of HIV (PMTCT) programs. BMC Pediatr. 2015 Feb 15;15:10. doi: 10.1186/s12887-015-0325-8. PMID 25886564
- [Result] Benki-Nugent S, Eshelman C, Wamalwa D, Langat A, Tapia K, Okinyi HM, John-Stewart G. Correlates of age at attainment of developmental milestones in HIV-infected infants receiving early antiretroviral therapy. Pediatr Infect Dis J. 2015 Jan;34(1):55-61. doi: 10.1097/INF.0000000000000526. PMID 25144793
- [Result] Slyker JA, Casper C, Tapia K, Richardson B, Bunts L, Huang ML, Wamalwa D, Benki-Nugent S, John-Stewart G. Accelerated suppression of primary Epstein-Barr virus infection in HIV-infected infants initiating lopinavir/ritonavir-based versus nevirapine-based combination antiretroviral therapy. Clin Infect Dis. 2014 May;58(9):1333-7. doi: 10.1093/cid/ciu088. Epub 2014 Feb 18. PMID 24550373
- [Result] Langat A, Benki-Nugent S, Wamalwa D, Tapia K, Ngugi E, Diener L, Richardson BA, Melvin A, John-Stewart GC. Lipid changes in Kenyan HIV-1-infected infants initiating highly active antiretroviral therapy by 1 year of age. Pediatr Infect Dis J. 2013 Jul;32(7):e298-304. doi: 10.1097/INF.0b013e31828afb2a. PMID 23385950
- [Derived] Benki-Nugent SF, Martopullo I, Laboso T, Tamasha N, Wamalwa DC, Tapia K, Langat A, Maleche-Obimbo E, Marra CM, Bangirana P, Boivin MJ, John-Stewart GC. High Plasma Soluble CD163 During Infancy Is a Marker for Neurocognitive Outcomes in Early-Treated HIV-Infected Children. J Acquir Immune Defic Syndr. 2019 May 1;81(1):102-109. doi: 10.1097/QAI.0000000000001979. PMID 30768490
- [Derived] Benki-Nugent S, Wamalwa D, Langat A, Tapia K, Adhiambo J, Chebet D, Okinyi HM, John-Stewart G. Comparison of developmental milestone attainment in early treated HIV-infected infants versus HIV-unexposed infants: a prospective cohort study. BMC Pediatr. 2017 Jan 17;17(1):24. doi: 10.1186/s12887-017-0776-1. PMID 28095807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were identified from Nairobi City Council clinics, the Kenyatta National Hospital (KNH) wards, and the HIV treatment clinic. Recruitment occurred from 2007-2009.
Pre-assignment Details: Of 140 infants enrolled, 37 infants died, 11 were lost, and 7 were withdrawn. Of 75 infants who completed 2 years ART pre-randomization, 33 were ineligible for randomization and 42 were randomized.
Groups:
- Continued HAART: After 24 months of HAART, infants were continued on HAART.
Period: Overall Study
Arm/Group | Continued HAART | Interrupted HAART
Started | 21 | 21
Completed | 18 | 21
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: following 24 months of HAART
Groups:
- Total: Total of all reporting groups
Arm/Group | Continued HAART | Interrupted HAART | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 29 [28.8 to 33.8] | 30.0 [29.3 to 34.9] | 30.0 [28.9 to 34.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  Kenya | 21 | 21 | 42
CD4% [Median (Inter-Quartile Range); unit: percent] | 33 [30 to 40] | 34 [32 to 38] | 33 [30 to 39]
Log10 HIV RNA level [Median (Inter-Quartile Range); unit: copies/ml] | 2.18 [2.18 to 2.64] | 2.18 [2.18 to 2.71] | 2.18 [2.18 to 2.71]

OUTCOME MEASURES:

1. Primary Outcome: Growth at 18 Months Post-randomization
Description: Weight and height will be transformed to the weight-for-age Z-score (i.e., WAZ) and height-for-age Z-score (i.e., HAZ) using World Health Organization Child Growth Standards, taking into account the infant's age and gender.
Time Frame: 18 months of post-randomization follow-up
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Continued HAART | Interrupted HAART
Number analyzed (Participants) | 21 | 21
z-score
  WAZ (z-score) | -0.57 [-0.88 to -0.28] | -0.17 [-0.56 to 0.37]
  HAZ (z-score) | -1.04 [-1.58 to -0.59] | -0.78 [-1.62 to 0]
Statistical Analysis 1: Comparison: Continued HAART vs Interrupted HAART; WAZ-score comparison at 18 months; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Continued HAART vs Interrupted HAART; HAZ score at 18 months; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Morbidity
Description: severe adverse events including death, pneumonia, diarrhea, and other adverse events
Time Frame: 18 months post-randomization
Measure: Number; unit: participants
Groups:
- Continue HAART: After 24 months of treatment with HAART, half the eligible infants will be randomized to continued treatment with HAART for 18 months.
Arm/Group | Continue HAART | Interrupted HAART
Number analyzed (Participants) | 21 | 21
participants
  Severe adverse events | 2 | 1
  Pneumonia | 4 | 3
  Diarrhea | 7 | 12
  Death | 1 | 0
Statistical Analysis 1: Comparison: Continue HAART vs Interrupted HAART; SAEs; Test type: Superiority or Other; p = 0.39, log rank or Cox regression; incidence with Cox regression utilized Anderson-Gill method to handle recurrent events
Statistical Analysis 2: Comparison: Continue HAART vs Interrupted HAART; Pneumonia; Test type: Superiority or Other; p = 0.60, Cox regression Anderson Gill
Statistical Analysis 3: Comparison: Continue HAART vs Interrupted HAART; Pneumonia; Test type: Superiority or Other; p = 0.60, Regression, Cox
Statistical Analysis 4: Comparison: Continue HAART vs Interrupted HAART; Diarrhea; Test type: Superiority or Other; p = 0.77, Regression, Cox
Statistical Analysis 5: Comparison: Continue HAART vs Interrupted HAART; Death; Test type: Superiority or Other; p = 0.29, Log Rank

ADVERSE EVENTS:
Time Frame: 18 months post-randomization
Arm/Group | Continued HAART | Interrupted HAART
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/21
Other Adverse Events (participants affected / at risk) | 21/21 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continued HAART (N=21) | Interrupted HAART (N=21)
Death (Infections and infestations) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continued HAART (N=21) | Interrupted HAART (N=21)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 21 | 20
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
High cholesterol (Metabolism and nutrition disorders) | 10 | 4
Diarrhea (Gastrointestinal disorders) | 7 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 14
Rash (Skin and subcutaneous tissue disorders) | 11 | 11
Anemia (Blood and lymphatic system disorders) | 12 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No